CLINICAL TRIAL: NCT01303380
Title: An Open-label, Multicenter, Efficacy and Safety Pilot Study of 6-month Canakinumab Treatment With up to 6-month Follow-up in Patients With Active Hyper-IgD Syndrome (HIDS)
Brief Title: Canakinumab in Patients With Active Hyper-IgD Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CACZ885D2402; 2010-020904-31 (EudraCT Number)
Record Dates: First submitted 2011-02-23; First posted 2011-02-24 (Estimated); Results first posted 2015-08-19 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-10

CONDITIONS: Mevalonate Kinase Deficiency
Keywords: Hyper IgD syndrome; canakinumab; HIDS; mevalonate kinase deficiency; MKD
MeSH Terms: conditions — Mevalonate Kinase Deficiency | interventions — canakinumab

ARMS (1):
- Canakinumab (Experimental)
  Interventions: Drug: Canakinumab

INTERVENTIONS:
Drug: Canakinumab

SUMMARY:
This pilot study is designed to evaluate the efficacy, the safety, and the pharmacokinetics (PK) / pharmacodynamics (PD) of canakinumab treatment in patients with HIDS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of HIDS proven by DNA analysis and/or enzymatic studies.
2. At time of start of drug treatment: active HIDS as evidenced by a physician global assessment of HIDS flare severity ≥ 2 and CRP values >10 mg/L (normal CRP < or = 10 mg/L).
3. Patients who have a history of > or = 3 febrile acute HIDS flares in a 6-month period when not receiving prophylaxis treatment (e.g. anakinra daily treatment) with a duration of each flare lasting > or = 4 days and limiting the normal daily activities.

Exclusion Criteria:

1. Pregnant or nursing (lactating) women.
2. History of being immunocompromised, including a positive HIV at screening (ELISA and Western blot) test result.
3. Positive Hepatitis B or Hepatitis C.
4. Live vaccinations within 3 months prior to the start of the trial
5. Positive tuberculosis screening test.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Spain (3):
  - Novartis Investigative Site, Esplugues de Llobregat, Barcelona
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Valencia, Valencia

REFERENCES:
- [Derived] Arostegui JI, Anton J, Calvo I, Robles A, Iglesias E, Lopez-Montesinos B, Banchereau R, Hong S, Joubert Y, Junge G, Pascual V, Yague J. Open-Label, Phase II Study to Assess the Efficacy and Safety of Canakinumab Treatment in Active Hyperimmunoglobulinemia D With Periodic Fever Syndrome. Arthritis Rheumatol. 2017 Aug;69(8):1679-1688. doi: 10.1002/art.40146. Epub 2017 Jul 5. PMID 28482144

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 3 centres in Spain.
Pre-assignment Details: A total of 10 participants were screened, 9 of which entered in the treatment period of the study, one participant was considered to be a screening failure.
Groups:
- Canakinumab: Participants received body weight stratified dosage of canakinumab (4 mg/kg for participants less than or equal to (≤) 40 kg or 300 mg for participants more than (>) 40 kg) as starting dose s.c. injection every 6 weeks during 6 months of treatment. The dose was escalated to additional 150 mg (2 mg/kg for participants ≤40 kg) dose at the moment of flare, and 450 mg (6 mg/kg for participants ≤40 kg) every 6 weeks, thereafter starting at Week 6 in participants who experienced a new Hyper-IgD with periodic fever syndrome (HIDS) flare between baseline and Week 4 as per investigator's discretion. If the flare occurred between Weeks 5-6, the participants received rescue medication and waited up to Week 6 to receive a total of 450 mg of canakinumab.
Period: Overall Study
Arm/Group | Canakinumab
Started | 9
Completed | 8
Not Completed | 1
Not completed — Lack of compliance to study procedures | 1

BASELINE CHARACTERISTICS:
Population: The analysis was performed in the Full Analysis Set (FAS), defined as all participants who received at least one application of study treatment and had at least one post-baseline assessment for primary efficacy variable.
Groups:
- Canakinumab: Participants received body weight stratified dosage of canakinumab (4 mg/kg for participants less than or equal to (≤) 40 kg or 300 mg for participants more than (>) 40 kg) as starting dose s.c. injection every 6 weeks during 6 months of treatment. The dose was escalated to additional 150 mg (2 mg/kg for participants ≤40 kg) dose at the moment of flare, and 450 mg (6 mg/kg for participants ≤40 kg) every 6 weeks, thereafter starting at Week 6 in participants who experienced a new HIDS flare between baseline and Week 4 as per investigator's discretion. If the flare occurred between Weeks 5-6, the participants received rescue medication and waited up to Week 6 to receive a total of 450 mg of canakinumab.
Arm/Group | Canakinumab
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: years] | 17.3 [5 to 29]
Age, Customized [Number; unit: participants]
  Children (2--11 years) | 3
  Adolescents (12--17 years) | 3
  Adults (18--64 years) | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Region of Enrollment [Number; unit: participants]
  Spain | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Flares Per Participant During Historical Period and Treatment Period
Description: A flare was defined as Physician Global Assessment of HIDS flare severity score of ≥ 2 and a C-reactive protein (CRP) value > 10 mg/L. Flares during a historical period were defined as most recent 6-months in which the participant has not received treatment for their HIDS other than symptomatic treatment with NSAIDs and/or corticosteroids.
Time Frame: Historical period, Month 6 (End of treatment period)
Population: The primary analysis was performed in the Full Analysis set (FAS) population defined as all participants who received at least one dose of study treatment and had at least one post baseline assessment.
Measure: Median (Full Range); unit: Number of flares
Arm/Group | Canakinumab
Number analyzed (Participants) | 9
Number of flares
  Historical period | 5 [3 to 12]
  Month 6 | 0 [0 to 2]

2. Secondary Outcome: Number of Flares Per Participant at During Treatment Period and 24 Month Extension Period
Description: A flare was defined as Physician Global Assessment of HIDS flare severity score of ≥ 2 and a CRP value > 10 mg/L.
Time Frame: Month 6 (End of treatment period), Month 36 (End of Long term treatment Period 2)
Population: The analysis was performed in the FAS population.
Measure: Median (Full Range); unit: Number of flares
Arm/Group | Canakinumab
Number analyzed (Participants) | 9
Number of flares
  Treatment period | 0 [0 to 2]
  Long term treatment period | 0 [0 to 1]

3. Secondary Outcome: Number of Participants Who Flared at Month 6, Month 24 and Month 36
Description: A flare was defined as Physician Global Assessment of HIDS flare severity score of ≥ 2 and a CRP value > 10 mg/L.
Time Frame: Baseline, Month 6 (End of treatment period), Month 24 (End of Long term treatment period 1) and Month 36 (End of Long term treatment period 2)
Population: The analysis was performed in the FAS population.
Measure: Number; unit: Number of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 9
Number of participants
  Treatment period | 2
  End of Long term treatment Period 1 | 4
  End of Long term treatment Period 2 | 2

4. Secondary Outcome: Number of Participants With Flare Events Based on Physician Assessed HIDS Flare Severity Score
Description: Physician global assessment of severity of HIDS after each flare was based on HIDS flare severity score, a 5- point scale: 0 = Absent signs/symptoms; 1 = Minimal signs/symptoms; 2 = Mild; 3= Moderate; 4 = Severe.
Time Frame: Any flare event [Baseline up to Month 36 (End of long term treatment period 2)]
Population: The analysis was performed in the FAS population. The 'n' signifies those participants evaluable for this measure at specified time points for each group, respectively.
Measure: Number; unit: Number of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 9
Number of participants
  Day 45, Absent (n=9) | 0
  Day 45, Minimal (n=9) | 0
  Day 45,Mild (n=9) | 0
  Day 45,Moderate (n=9) | 1
  Day 45,Severe (n=9) | 0
  Flare/Unscheduled visit 1, Absent (n=2) | 2
  Flare/Unscheduled visit 1, Minimal (n=2) | 0
  Flare/Unscheduled visit 1, Mild (n=2) | 1
  Flare/Unscheduled visit 1, Moderated (n=2) | 1
  Flare/Unscheduled visit 1, Severe (n=2) | 0
  Flare/Unscheduled visit 2, Absent (n=2) | 1
  Flare/Unscheduled visit 2, Minimal (n=2) | 0
  Flare/Unscheduled visit 2, Mild (n=2) | 1
  Flare/Unscheduled visit 2, Moderate (n=2) | 0
  Flare/Unscheduled visit 2, Severe (n=2) | 0
  Flare/Unscheduled visit 3, Absent (n=2) | 1
  Flare/Unscheduled visit 3, Minimal (n=2) | 0
  Flare/Unscheduled visit 3, Mild (n=2) | 0
  Flare/Unscheduled visit 3, Moderate (n=2) | 1
  Flare/Unscheduled visit 3, Severe (n=2) | 0
  End of Treatment period, Absent (n=7) | 0
  End of Treatment period, Minimal (n=7) | 0
  End of Treatment period, Mild (n=7) | 4
  End of Treatment period, Moderate (n=7) | 3
  End of Treatment period, Severe (n=7) | 0
  End of Follow-up period, Absent (n=8) | 0
  End of Follow-up period, Minimal (n=8) | 1
  End of Follow-up period, Mild (n=8) | 0
  End of Follow-up period, Moderate (n=8) | 0
  End of Follow-up period, Severe (n=8) | 0
  Long term period 1, Flare 1, Absent (n=3) | 0
  Long term period 1, Flare 1, Minimal (n=3) | 1
  Long term period 1, Flare 1, Mild (n=3) | 1
  Long-term 12 M period, Flare 1, Moderate (n=3) | 1
  Long-term 12 M period, Flare 1, Severe (n=3) | 0
  Long term period 1, Flare 2, Absent (n=1) | 0
  Long-term 12 M period, Flare 2, Minimal (n=1) | 0
  Long-term 12 M period, Flare 2, Mild (n=1) | 1
  Long term period 1, Flare 2, Moderate (n=1) | 0
  Long term period 1, Flare 2, Severe (n=1) | 0
  Long term period 1, Flare 3, Absent (n=1) | 0
  Long term period 1, Flare 3, Minimal (n=1) | 0
  Long term period 1, Flare 3, Mild (n=1) | 1
  Long term period 1, Flare 3, Moderate (n=1) | 0
  Long term period 1, Flare 3, Severe (n=1) | 0
  Long term period 2, Absent (n=2) | 1
  Long term period 2, Minimal (n=2) | 0
  Long term period 2, Mild (n=2) | 1
  Long term period 2, Moderate (n=2) | 0
  Long term period 2, Severe (n=2) | 0

5. Secondary Outcome: Number of Participants With Flare Events Based on Participant Assessed HIDS Flare Severity Score
Description: Participant's global assessment of severity of HIDS after each flare was based on HIDS flare severity score, a 5-point scale: 0 = Absent signs/symptoms; 1 = Minimal signs/symptoms; 2 = Mild; 3= Moderate; 4 = Severe. Same investigator assessed the same participant throughout the study to ensure consistency between assessments. Investigators reviewed every participant's diary at each visit after their own clinical assessment.
Time Frame: Baseline, Month 6 (End of treatment period), Month 12 (End of follow up period), Month 24 (End of Long term treatment period 1) and Month 36 (End of Long term treatment period 2)
Population: The analysis was performed in the FAS population.
Measure: Number; unit: Number of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 9
Number of participants
  Treatment period, Absent | 0
  Treatment period, Minimal | 0
  Treatment period, Mild | 1
  Treatment period, Moderate | 1
  Treatment period, Severe | 0
  Follow-up period, Absent | 0
  Follow-up period, Minimal | 0
  Follow-up period, Mild | 0
  Follow-up period, Moderate | 2
  Follow-up period, Severe | 0
  Long term period 1, Absent | 0
  Long term period 1, Minimal | 1
  Long term period 1, Mild | 1
  Long term period 1, Moderate | 2
  Long term period 1, Severe | 0
  Long term period 2, Absent | 0
  Long term period 2, Minimal | 1
  Long term period 2, Mild | 0
  Long term period 2, Moderate | 0
  Long term period 2, Severe | 0

6. Secondary Outcome: Percentage of Participants With Defined Grades of Participants Assessed Symptom Control
Description: Participants were assessed by participants/parent (participants aged 6-18 years) for control of signs and symptoms associated with HIDS based on 5-point scale: 0 = No control; 1 = Poor control; 2 = Somewhat control; 3 = Good control; and 4= Excellent control.
Time Frame: as for outcome 5
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 9
Percentage of participants
  Treatment period, No control (n=9) | 0
  Treatment period, Poor control (n=9) | 0
  Treatment period, Somewhat control (n=9) | 11.11
  Treatment period, Good control (n=9) | 33.33
  Treatment period, Excellent control (n=9) | 55.56
  Follow-up period, No control (n=9) | 0
  Follow-up period, Poor control (n=9) | 0
  Follow-up period, Somewhat control (n=9) | 0
  Follow-up period, Good control (n=9) | 33.33
  Follow-up period, Excellent control (n=9) | 66.67
  Long term period 1, No control (n=8) | 0
  Long term period 1, Poor control (n=8) | 0
  Long term period 1, Somewhat control (n=8) | 12.5
  Long term period 1, Good control (n=8) | 25
  Long term period 1, Excellent control (n=8) | 62.5
  Long term period 2, No control (n=8) | 0
  Long term period 2, Poor control (n=8) | 0
  Long term period 2, Somewhat control (n=8) | 0
  Long term period 2, Good control (n=8) | 12.5
  Long term period 2, Excellent control (n=8 | 87.5

7. Secondary Outcome: Percentage of Participants With Defined Grades of Physician Assessed Symptom Control
Description: Participants were assessed by physician for control of signs and symptoms associated with HIDS based on 5-point scale: 0 = No control; 1 = Poor control; 2 = Somewhat control; 3 = Good control; and 4= Excellent control.
Time Frame: as for outcome 5
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 9
Percentage of participants
  Treatment period, No control (n=9) | 0
  Treatment period, Poor control (n=9) | 0
  Treatment period, Somewhat control (n=9) | 0
  Treatment period, Good control (n=9) | 44.44
  Treatment period, Excellent control (n=9) | 55.56
  Follow-up period, No control (n=9) | 0
  Follow-up period, Poor control (n=9) | 0
  Follow-up period, Somewhat control (n=9) | 0
  Follow-up period, Good control (n=9) | 33.33
  Follow-up period, Excellent control (n=9) | 66.67
  Long term period 1, No control (n=8) | 0
  Long term period 1, Poor control (n=8) | 0
  Long term period 1, Somewhat control (n=8) | 12.5
  Long term period 1, Good control (n=8) | 25
  Long term period 1, Excellent control (n=8) | 62.5
  Long term period 2, No control (n=8) | 0
  Long term period 2, Poor control (n=8) | 0
  Long term period 2, Somewhat control (n=8) | 0
  Long term period 2, Good control (n=8) | 0
  Long term period 2, Excellent control (n=8 | 100

8. Secondary Outcome: Percentage of Participants Experiencing Fever as Assessed by Physician's Global Assessment
Description: Fever severity was assessed by physician after each flare using a 5-point scale: 0 =Absent signs/symptoms; 1 = Minimal signs/symptoms; 2 = Mild; 3 = Moderate; 4 = Severe.
Time Frame: as for outcome 5
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 9
Percentage of participants
  Treatment period, Absent (n=9) | 88.89
  Treatment period, Minimal (n=9) | 11.11
  Treatment period, Mild (n=9) | 0
  Treatment period, Moderate (n=9) | 0
  Treatment period, Severe (n=9) | 0
  Follow-up period, Absent (n=9) | 100
  Follow-up period, Minimal (n=9) | 0
  Follow-up period, Mild (n=9) | 0
  Follow-up period, Moderate (n=9) | 0
  Follow-up period, Severe (n=9) | 0
  Long term period 1, Absent (n=8) | 75
  Long term period 1, Minimal (n=8) | 12.5
  Long term period 1, Mild (n=8) | 12.5
  Long term period 1, Moderate (n=8) | 0
  Long term period 1, Severe (n=8) | 0
  Long term period 2, Absent (n=8) | 100
  Long term period 2, Minimal (n=8) | 0
  Long term period 2, Mild (n=8) | 0
  Long term period 2, Moderate (n=8) | 0
  Long term period 2, Severe (n=8) | 0

9. Secondary Outcome: Percentage of Participants Experiencing Apthus Ulcers as Assessed by Physician's Global Assessment
Description: Apthus ulcers were assessed by physician after each flare using a 5-point scale: 0 =Absent signs/symptoms; 1 = Minimal signs/symptoms; 2 = Mild; 3 = Moderate; 4 = Severe.
Time Frame: as for outcome 5
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 9
Percentage of participants
  Treatment period, Absent (n=9) | 88.89
  Treatment period, Minimal (n=9) | 0
  Treatment period, Mild (n=9) | 11.11
  Treatment period, Moderate (n=9) | 0
  Treatment period, Severe (n=9) | 0
  Follow-up period, Absent (n=9) | 100
  Follow-up period, Minimal (n=9) | 0
  Follow-up period, Mild (n=9) | 0
  Follow-up period, Moderate (n=9) | 0
  Follow-up period, Severe (n=9) | 0
  Long term period 1, Absent (n=8) | 100
  Long term period 1, Minimal (n=8) | 0
  Long term period 1, Mild (n=8) | 0
  Long term period 1, Moderate (n=8) | 0
  Long term period 1, Severe (n=8) | 0
  Long term period 2, Absent (n=8) | 100
  Long term period 2, Minimal (n=8) | 0
  Long term period 2, Mild (n=8) | 0
  Long term period 2, Moderate (n=8) | 0
  Long term period 2, Severe (n=8) | 0

10. Secondary Outcome: Percentage of Participants Experiencing Lymphadenopathy as Assessed by Physician's Global Assessment
Description: Lymphadenopathy severity was assessed by physician after each flare using a 5-point scale: 0 =Absent signs/symptoms; 1 = Minimal signs/symptoms; 2 = Mild; 3 = Moderate; 4 = Severe.
Time Frame: as for outcome 5
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 9
Percentage of participants
  Treatment period, Absent (n=9) | 88.89
  Treatment period, Minimal (n=9) | 11.11
  Treatment period, Mild (n=9) | 0
  Treatment period, Moderate (n=9) | 0
  Treatment period, Severe (n=9) | 0
  Follow-up period, Absent (n=9) | 77.78
  Follow-up period, Minimal (n=9) | 22.22
  Follow-up period, Mild (n=9) | 0
  Follow-up period, Moderate (n=9) | 0
  Follow-up period, Severe (n=9) | 0
  Long term period 1, Absent (n=8) | 87.5
  Long term period 1, Minimal (n=8) | 12.5
  Long term period 1, Mild (n=8) | 0
  Long term period 1, Moderate (n=8) | 0
  Long term period 1, Severe (n=8) | 0
  Long term period 2, Absent (n=8) | 100
  Long term period 2, Minimal (n=8) | 0
  Long term period 2, Mild (n=8) | 0
  Long term period 2, Moderate (n=8) | 0
  Long term period 2, Severe (n=8) | 0

11. Secondary Outcome: Percentage of Participants Experiencing Abdominal Pain as Assessed by Physician's Global Assessment
Description: Abdominal pain was assessed by physician after each flare using a 5-point scale: 0 =Absent signs/symptoms; 1 = Minimal signs/symptoms; 2 = Mild; 3 = Moderate; 4 = Severe.
Time Frame: as for outcome 5
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 9
Percentage of participants
  Treatment period, Absent (n=9) | 100
  Treatment period, Minimal (n=9) | 0
  Treatment period, Mild (n=9) | 0
  Treatment period, Moderate (n=9) | 0
  Treatment period, Severe (n=9) | 0
  Follow-up period, Absent (n=9) | 100
  Follow-up period, Minimal (n=9) | 0
  Follow-up period, Mild (n=9) | 0
  Follow-up period, Moderate (n=9) | 0
  Follow-up period, Severe (n=9) | 0
  Long term period 1, Absent (n=8) | 87.5
  Long term period 1, Minimal (n=8) | 12.5
  Long term period 1, Mild (n=8) | 0
  Long term period 1, Moderate (n=8) | 0
  Long term period 1, Severe (n=8) | 0
  Long term period 2, Absent (n=8) | 100
  Long term period 2, Minimal (n=8) | 0
  Long term period 2, Mild (n=8) | 0
  Long term period 2, Moderate (n=8) | 0
  Long term period 2, Severe (n=8) | 0

12. Secondary Outcome: Time to Resolution of the Initial Flare After First Canakinumab Treatment
Description: Time to resolution of the initial flare after first dose of canakinumab was determined.
Time Frame: Day 1 (Baseline), Day 28
Population: The analysis was performed in the FAS population.
Measure: Median (Full Range); unit: Days
Arm/Group | Canakinumab
Number analyzed (Participants) | 9
Days | 3 [1 to 5]

13. Secondary Outcome: Change From Baseline in Inflammation Markers Over Time up to Month 24
Description: The C-reactive Protein (CRP) and/or Serum amyloid A protein (SAA) were used as inflammatory markers. The normal range of CRP was 0-10 mg/L.
Time Frame: as for outcome 5
Population: The analysis was performed in the FAS population. The 'n' signifies those participants evaluable for this measure at specified time points for each group respectively.
Measure: Median (Full Range); unit: milligram(s)/liter
Arm/Group | Canakinumab
Number analyzed (Participants) | 9
milligram(s)/liter
  CRP- 6 month (Treatment period), (n=6) | -120.5 [-164 to -23]
  CRP- 6 month (Follow-up period), (n=9) | -111 [-164 to -23]
  CRP- Long term period 1, (n=8) | -113.55 [-159.5 to -49.9]
  CRP- Long term period 2, (n=8) | -125.2 [-164 to -34.1]
  SAA- 6 month (Treatment period), (n=1) | -624.2 [-624.2 to -23]
  SAA- 6 month (Follow-up period), (n=2) | -685.95 [-748.2 to -623.7]
  SAA- Long term period 1, (n=2) | -684.1 [-749.2 to -619]
  SAA- Long term period 2, (n=2) | -686.7 [-747.7 to -625.7]

14. Secondary Outcome: Health Assessment Questionnaire (HAQ) Global Score in Adults Over Time
Description: Participants were assessed for health-related quality of life (HRQoL) based on Health Assessment Questionnaire (HAQ). HAQ was an eight 8 categories questionnaire representing all activities related to physical function. Each category has various sub-categories, which were rated by the participants on a 4- point difficulty scale: 0 = any difficulty; 1 = some difficulty; 2 = much difficulty; 3 = unable to do. The total score was the mean of the 8 scores, and ranged from 0 (no disability) to 3 (completely disabled).
Time Frame: as for outcome 5
Population: The analysis was performed in the FAS population. The 'n' signifies those participants evaluable for this measure at specified time points for each group respectively. Here "Number of participants analyzed" signifies the participants assessed for HAQ during study.
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Canakinumab
Number analyzed (Participants) | 6
Score on a scale
  Treatment period, (n=3) | 0 [0 to 0]
  Follow-up period, (n=4) | 0 [0 to 0]
  Long term period 1, (n=5) | 0 [0 to 1]
  Long term period 2, (n=4) | 0 [0 to 0]

15. Secondary Outcome: Childhood Health Assessment Questionnaire (CHAQ) Global Score in Children Over Time
Description: Participants or their parents (participants aged 6 to 17 years) were assessed for HRQoL based on Childhood Health Assessment Questionnaire (CHAQ). CHAQ was an eight domain questionnaire representing functional capacity and independence, evaluated for previous week. Each domain was rated on a 4-point difficulty scale: 0 = any difficulty; 1 = some difficulty; 2 = much difficulty; 3 = unable to do.The total score is the mean from the 8 scores, and ranges from 0 (no disability) to 3 (completely disabled).
Time Frame: as for outcome 5
Population: The analysis was performed in the FAS population. The 'n' signifies those participants evaluable for this measure at specified time points for each group respectively. Here "Number of participants analyzed" signifies the participants assessed for CHAQ during study.
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Canakinumab
Number analyzed (Participants) | 6
Score on a scale
  End to treatment period (n= 2) | 0 [0 to 0]
  End to follow-up period (n=4) | 0.1 [0 to 1]
  Long term period 1, (n=2) | 0.1 [0 to 1]
  Long term period 2, (n=1) | 0.1 [0 to 1]

16. Secondary Outcome: Percentage of Participants Who Received Dose Up-titration During 6-month Treatment Period
Description: Participants who experienced a new HIDS flare between baseline and Week 4 and received an escalated dose of 450 mg of canakinumab every 6 weeks thereafter starting at Week 6 were determined.
Time Frame: Day 1 up to Month 6 (End of follow up)
Population: The analysis was performed in the FAS population.
Measure: Number; unit: Percentage of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 9
Percentage of participants | 22.22

17. Secondary Outcome: Duration of Flares Experienced During the Study
Description: Flare was defined as Physician Global Assessment of HIDS flare severity score of ≥ 2 and a CRP value > 10 mg/L. The change in post canakinumab treatment flare duration during the study were assessed as compared to historical period.
Time Frame: as for outcome 5
Population: as for outcome 13
Measure: Median (Full Range); unit: Days
Arm/Group | Canakinumab
Number analyzed (Participants) | 9
Days
  Treatment period, (n=3) | 3 [2 to 4]
  Follow-up period, (n=7) | 4 [2 to 10]
  Long term period 1, (n=6) | 3.5 [2 to 8]
  Long term period 2, (n=2) | 8.5 [6 to 11]

18. Secondary Outcome: Time to Flare After the Last Dose of Canakinumab During the Follow-up Period
Description: The median time to flare by the participants after administration of the last dose of canakinumab during the follow-up period was analysed using Kaplan-Meier method.
Time Frame: Last dose of canakinumab treatment in follow-up period to end of follow-up period (Day 337)
Population: The analysis was performed on the FAS population. Here "Number of participants analysed" signifies the participants assessed for time to flare after the last dose of canakinumab during follow-up period.
Measure: Median (Full Range); unit: days
Arm/Group | Canakinumab
Number analyzed (Participants) | 7
days | 110 [62 to 196]

19. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Adverse events (AEs) were defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. Serious adverse events (SAEs) were defined as any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalisation, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgement of investigators represent significant hazards.
Time Frame: Day 1 (Start of study treatment) up to Month 36 (End of study)
Population: The analysis was performed on Safety Set (SAF) population defined as all participants who received at least one application of study treatment and had at least one post-baseline safety assessment.
Measure: Number; unit: Number of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 9
Number of participants
  Adverse events | 9
  Serious adverse events | 4

20. Secondary Outcome: Participants Who Received Rescue Treatment
Description: Participants who experienced flares were treated with corticosteroids and NSAIDs as rescue medication.
Time Frame: Baseline up to Month 36 (End of study)
Population: The analysis was performed on the FAS population.
Measure: Number; unit: Percentage of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 9
Percentage of participants | 11.11

21. Secondary Outcome: Serum Concentration-time Profile of Canakinumab
Description: Canakinumab concentrations in serum were assessed for evaluating pharmacokinetics (PK) of the drug.
Time Frame: Day 1 (Pre-dose), Day 4, Day 15, Day 43, Day 85, Day 127, Day 169 (End of treatment period), Day 197, Day 225, Day 253, Day 281, Day 309, and Day 337 (End of follow-up period) (Post-dose)
Population: The analysis was performed on the FAS population.
Measure: Mean (Standard Deviation); unit: microgram(s)/milliliter
Arm/Group | Canakinumab
Number analyzed (Participants) | 9
microgram(s)/milliliter
  Day 4 | 28.8 (7.9)
  Day 15 | 26.9 (8)
  Day 43 | 12.7 (4.6)
  Day 85 | 19.4 (9.6)
  Day 127 | 23.8 (12.8)
  Day 169 | 24 (13.4)
  Day 197 | 12.6 (13.7)
  Day 225 | 11.5 (7.9)
  Day 253 | 6.5 (4.8)
  Day 281 | 1.6 (1.6)
  Day 309 | 0.9 (1)
  Day 337 | 32.6 (15.9)

22. Secondary Outcome: Serum Concentration of Total Interleukin-1β Antibody (IL-1β)
Description: Pharmacodynamics of canakinumab was assessed by total IL-1β (sum of free and bound canakinumab) concentration, determined in serum by means of sandwich ELISA assay with limit of detection at 0.1 picogram/millilitre.
Time Frame: as for outcome 21
Population: The analysis was performed on the FAS population.
Measure: Mean (Standard Deviation); unit: picogram(s)/milliliter
Arm/Group | Canakinumab
Number analyzed (Participants) | 9
picogram(s)/milliliter
  Day 4 | 27.3 (25.2)
  Day 15 | 22.2 (14.7)
  Day 43 | 21.8 (13.9)
  Day 85 | 27.3 (14)
  Day 127 | 24.3 (12.1)
  Day 169 | 32.5 (17.9)
  Day 197 | 16.3 (5.9)
  Day 225 | 17 (8.3)
  Day 253 | 10.2 (5.8)
  Day 281 | 4.9 (3.3)
  Day 309 | 3.7 (2)
  Day 337 | 49.1 (60.2)

23. Secondary Outcome: Number of Participants Exhibiting Anti-canakinumab Antibodies at Any Visit
Description: Immunogenicity assessment included determination of anti-canakinumab (ACZ885) antibodies in serum samples using bridging ECLIA assay.
Time Frame: Baseline up to Month 36 (End of study)
Population: The analysis was performed on the FAS population.
Measure: Number; unit: Number of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 9
Number of participants | 0

ADVERSE EVENTS:
Time Frame: Serious Adverse Events are monitored from date of First Participant First Visit (FPFV) until Last Participant Last Visit (LPLV). All other adverse events are monitored from First Participant First Treatment until LPLV.
Arm/Group | Canakinumab
Serious Adverse Events (participants affected / at risk) | 4/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab (N=9)
Anaemia (Blood and lymphatic system disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 1
Cellulitis (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Streptococcal bacteraemia (Infections and infestations) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab (N=9)
Tachycardia (Cardiac disorders) | 1
Conjunctival hyperaemia (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Aphthous stomatitis (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Impaired healing (General disorders) | 1
Influenza like illness (General disorders) | 1
Pyrexia (General disorders) | 4
Bronchitis (Infections and infestations) | 1
Candidiasis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Impetigo (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Pharyngotonsillitis (Infections and infestations) | 3
Respiratory tract infection (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Tonsillitis streptococcal (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Vulvovaginal mycotic infection (Infections and infestations) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Scoliosis (Musculoskeletal and connective tissue disorders) | 1
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Vaginal ulceration (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 1
Tooth extraction (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (i.e, data from all sites) in the clinical trial.